CLINICAL TRIAL: NCT03891498
Title: The Effect of Loading Dose of Magnesium Sulfate on Uterine, Umbilical, and Fetal Middle Cerebral Arteries Doppler, Biophysical Profile, CTG, Maternal Vital Signs in Women With Severe Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 53
Record Dates: First submitted 2019-03-24; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MgSO4 (Experimental): The magnesium sulfate will be given according to the regimen of 6 grams intravenous over 20 minutes as a loading dose.
  Interventions: Drug: MgSO4

INTERVENTIONS:
Drug: MgSO4 — The magnesium sulfate will be given according to the regimen of 6 grams intravenous over 20 minutes as a loading dose.

SUMMARY:
100 women with severe preeclanpsia received Magnesium sulfate 6 grams intravenous over 20 minutes as a loading dose. Resistance index [RI], pulsatility index [PI] and systolic/diastolic [S/D] ratio of the umbilical artery, uterine aryery and fetal middle cerebral artery before and repeated 20 minutes after intravenous administration of 6 grams of magnesium sulphate (loading dose) over 20 minutes . fetal breathing movements and fetal gross movements are counted within 20 minutes, before and after intravenous administration of 6 grams of magnesium sulphate (loading dose) over 20 minutes

DETAILED DESCRIPTION:
100 women with severe preeclanpsia received Magnesium sulfate 6 grams intravenous over 20 minutes as a loading dose. Resistance index [RI], pulsatility index [PI] and systolic/diastolic [S/D] ratio of the umbilical artery, uterine aryery and fetal middle cerebral artery before and repeated 20 minutes after intravenous administration of 6 grams of magnesium sulphate (loading dose) over 20 minutes . fetal breathing movements and fetal gross movements are counted within 20 minutes, before and after intravenous administration of 6 grams of magnesium sulphate (loading dose) over 20 minutes

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Primigravida or Multigravida.
* Pregnant females ≥ 37 weeks of gestation.
* Diagnosed as severe preeclampsia by the following criteria:

  * Sustained systolic blood pressure of ≥160 mmHg or a sustained diastolic blood pressure of ≥ 110 mmHg.
  * Proteinuria measured as +1 or more by dipstick or 24 hours urine collection with proteinuria ≥ 0.3 grams.
  * Oliguria or creatinine > 1.1 mg%.
  * Laboratory findings characteristic of HELLP syndrome.
  * Symptoms suggestive of severe preeclampsia ; severe headache, blurring of vision, epigastric pain.

Exclusion Criteria:

* Multifetal pregnancy.
* History of epilepsy.
* Patients with diabetes.
* Patients with renal disease.
* Fetuses with congenital anomalies.
* Patients receiving anticoagulants e.g. heparin (unfractionated or low molecular weight).
* Patients with severe IUGR.
* Patients with accidental hemorrhage.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in uterine artery resistance index | 15 minutes after the loading dose of MgSO4
  Doppler assessment of uterine artey RI

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt